CLINICAL TRIAL: NCT01461174
Title: Effects of 15-day Donepezil and Memantine on Cognitive Functions After a 24 Hours Sleep Deprivation Challenge in Healthy Volunteers: a Double-blind, Placebo-controlled, Randomised, Cross-over Study, With Modafinil as Positive Control
Brief Title: Effects of Donepezil and Memantine on Cognitive Functions After a Sleep Deprivation Challenge in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qualissima (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: WP1P001; 2011-000344-25 (EudraCT Number)
Record Dates: First submitted 2011-10-17; First posted 2011-10-27 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
Keywords: Sleep deprivation; Cognitive Functions; young male
MeSH Terms: conditions — Sleep Deprivation | interventions — Modafinil; Donepezil; Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Modafinil (Experimental): 200 mg tablet, single dose
  Interventions: Drug: Modafinil
- Donepezil (Experimental): 5 mg tablet one per day, 15 days
  Interventions: Drug: Donepezil
- Memantine (Experimental): 10 mg tablet one per day, 15 days
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Modafinil — 200 mg tablet, single dose
  Arms: Modafinil
Drug: Donepezil — Donepezil or placebo, 5 mg tablet one per day, 15 days
  Arms: Donepezil
Drug: Memantine — Memantine or placebo, 10 mg tablet one per day, 15 days
  Arms: Memantine

SUMMARY:
The aim of this study is to assess the utility of sleep deprivation as a potential model for prediction of clinical efficacy using a combination of cognitive physiological endpoints.

DETAILED DESCRIPTION:
BACKGROUND:

With the inherent difficulty of detecting significant improvements in cognitive performance in normal healthy subjects, it is presently incredibly hard to predict and select efficacious agents early in the drug development process. As such the potential success of novel therapeutic agents for the symptomatic relief of Alzheimer's disease (AD) is largely unknown until the drugs enter relatively large studies, assessing clinical outcome over at least a six month period. To try to overcome this issue, clinical scientists have focused their attention to the development of cognitive endpoints/biomarkers that can be detected in a number of experimental paradigms where cognitive impairments akin to those observed in AD, have been artificially induced.Based on the scientific literature, the use of total Sleep Deprivation in healthy volunteers seems to be a good paradigm to assess potential anti-AD agents.

It is the first multicenter study that combines 3 complementary approaches via a standardization of the sleep deprivation model: cognitive evaluations, imaging and neurophysiology.

STUDY OBJECTIVE(S)

Primary:

The study aim is to assess the utility of sleep deprivation as a potential model for prediction of clinical efficacy using a combination of cognitive physiological endpoints.

The main goals are to test the effects of donepezil and memantine treatment on cognitive functions in young healthy deprived subjects and to assess the potential restoring effect of the two drugs on cognitive functions induce by sleep deprivation.

Secondary:

* To assess that Sleep Deprivation model results in cognitive impairments
* To determine the sensitivity of the model by testing the restoring effects of one single dose of modafinil
* To investigate the reversal effect of modafinil on EEG under sleep deprivation.
* To investigate the reversal effect of modafinil on fMRI acquisitions under sleep deprivation (subjects that will be included in Toulouse will not have fMRI)
* To investigate the influence of donepezil and memantine on EEG under sleep deprivation.
* To investigate the influence of donepezil and memantine on fMRI acquisitions under sleep deprivation (subjects that will be included in Toulouse will not have fMRI).

STUDY DESIGN The study is a phase I, multicentric (Lille, Marseille, Toulouse), randomised, placebo-controlled, cross-over design.

STUDY POPULATION Healthy young male subjects from 25 to 40 years-old (36 subjects randomized)

PRIMARY ENDPOINT(S) AND MAIN SECONDARY ENDPOINT(S)

Primary endpoint:

N-back test

Secondary endpoints:

* Other cognitive assessments
* Imaging
* Neurophysiology

ELIGIBILITY:
Inclusion Criteria:

Demography

1. Healthy male subjects aged between 25 and 40 years-old inclusive
2. BMI between 18 kg/m2 to 27 kg/m2

   Health status
3. The subjects is in good health on the basis of the medical interview (medical history, symptoms) and the physical examination, vital signs and the results of blood chemistry and hematology.
4. ECG (12 leads) normal (120 < PR < 200 ms; QRS < 120ms; QTcF < 450ms) and/or without clinically relevant impairments as judged by investigator.
5. The subject does not smoke or smokes a maximum of 5 cigarettes per day and is able to stop during the days of the study.
6. No claustrophobia (fMRI)
7. The subject has normal visual and auditory abilities

   Specific to the study
8. Habitual good sleeping: sleeping on average 6,5 to 9 hours each night in the past month assessed by the Pittsburgh Quality Index.
9. Regular sleeping hours whereby they sleep no later than 1 am and rise before 9 am in the past month assessed by the Pittsburgh Quality Index.
10. The subject can complete the neuropsychological test battery during the training session
11. The subject corresponds to an extravert personality according to the Eysenck Personality Inventory
12. The subject is right-handed (Edinburgh Handedness Inventory, Imaging measurement condition).

    Regulations
13. The subjects is able to read and understand the Information Form and comply with the protocol instructions and restrictions
14. Subjects are covered by a social insurance
15. Subjects have provided written informed consent

Exclusion Criteria:

Medical history and clinical status

1. History or presence of psychiatric illness assessed by a psychiatric interview with the Mini-International Neuropsychiatric Interview (M.I.N.I-DSM IV).
2. History or presence of neurologic illness or others illnesses (general medical interview)
3. The subject has caffeine intake of greater than 5 drinks per day or excessive energy drink type intake.
4. The subject has an orthostatic blood pressure reduction > 20 mm Hg, based on a difference of systolic blood pressure between supine and after standing for 3 minutes.

   General conditions
5. The patient, in the opinion of the investigator, is unlikely to comply with the study protocol or is unsuitable for any other reason
6. The subject participates to another clinical trial or is still being within a washout period of a previous clinical trial, or subjects who received more than 4500 euros in the previous 12 months.

   Specific to the study
7. History or presence of daytime sleepiness with the Epworth scale (score > 10, pathological sleepiness).
8. History of obstructive sleep apnea assessed by the Berlin questionnaire.
9. History of periodic leg movements assessed by Restless Legs Syndrome questionnaire.
10. Extreme chronotypes: score at the Horne Ostberg scale (< 31 or > 69).
11. Jet lag > 2 hours in the last two weeks.
12. No time-shifted work during the last month.

Ages: 25 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in N-back | Day 1 and Day 2 for each of the 5 Period
  The N-back test is both sensitive to SD in healthy volunteers and this test belongs to ADNI cognitive battery which is validated in Alzheimer's disease patients,considered as primary endpoint.

SECONDARY OUTCOMES:
Other cognitive assessments | Day 1 and Day 2 for each of the 5 Period
  CANTAB Battery, Memory Rey Auditory Verbal Learning Test (AVLT), Digit Span Test, Verbal Fluency task
fMRI | Day 1 and Day 2 for each of the 5 Period
  Resting fMRI, fMRI Memory task
Rest-EEG and P300 after auditory-ball paradigm Rest-EEG and P300 after auditory-ball paradigm Rest-EEG and P300 after auditory-ball paradigm | Day 1 and Day 2 for each of the 5 Period
  Rest-EEG and P300 after auditory-ball paradigm

CONTACTS AND LOCATIONS:
Overall Officials: Christine Audebert, Principal Investigator — CIC CPCET
Locations (2):
- France (2):
  - CIC, Lille
  - MEDES, Toulouse